CLINICAL TRIAL: NCT02698683
Title: Lymphocyte Count as a Sign of Immunoparalysis and Its Correlation With Nutritional Status in Septic Pediatric Intensive Care Patients: A Pilot Study
Brief Title: Lymphocyte Count as a Sign of Immunoparalysis and Its Correlation With Nutritional Status in Septic Pediatric Patients
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Talita Freitas Manzoli, Medical doctor, University of Sao Paulo
Other Study IDs: 2015-LCSINS
Record Dates: First submitted 2016-02-22; First posted 2016-03-04 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-02

CONDITIONS: Lymphopenia
Keywords: Nutrition; Lymphocyte Count; Immunoparalysis; nutritional status of septic patients
MeSH Terms: conditions — Lymphopenia | interventions — Lymphocyte Count

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- malnourished: low zinc, low albumin, anthropometric measures lower than percentile 5 lymphocyte count
  Interventions: Other: lymphocyte count
- well nourished: normal zinc, normal albumin, anthropometric measures higher than percentile 5 lymphocyte count
  Interventions: Other: lymphocyte count

INTERVENTIONS:
Other: lymphocyte count — lymphocyte count

SUMMARY:
Participants were classified as normal or malnourished according to anthropometric measures. Serum albumin and zinc were recovered on the 1st and 7th days of hospitalization. Lymphocyte count was also recorded on the 1st and 7th days.

DETAILED DESCRIPTION:
The investigators enrolled 14 consecutive patients with sepsis. Patients were classified as normal or malnourished according to anthropometric measures. As an additional evaluation of nutritional status, serum albumin and zinc were recovered on the 1st and 7th days of hospitalization. Lymphocyte count was also recorded on the 1st and 7th days. Investigators correlated nutritional status with lymphocyte count and zinc dosage.

ELIGIBILITY:
Inclusion Criteria:

* septic patients

Exclusion Criteria:

-

Ages: 1 Month to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: pediatric septic patients
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2014-02; Primary Completion 2015-06 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
presence of lymphopenia | seven days

IPD SHARING:
Plan to Share IPD: No
there is no plan to share data

REFERENCES:
- [Result] Delgado AF, Okay TS, Leone C, Nichols B, Del Negro GM, Vaz FA. Hospital malnutrition and inflammatory response in critically ill children and adolescents admitted to a tertiary intensive care unit. Clinics (Sao Paulo). 2008 Jun;63(3):357-62. doi: 10.1590/s1807-59322008000300012. PMID 18568246
- [Derived] Manzoli TF, Delgado AF, Troster EJ, de Carvalho WB, Antunes AC, Marques DM, Zamberlan P. Lymphocyte count as a sign of immunoparalysis and its correlation with nutritional status in pediatric intensive care patients with sepsis: A pilot study. Clinics (Sao Paulo). 2016 Nov 1;71(11):644-649. doi: 10.6061/clinics/2016(11)05. PMID 27982165